CLINICAL TRIAL: NCT06867757
Title: Targeted Realtime Assessment of Chronic Pain (TRAC-Pain) in Youth
Brief Title: Targeted Realtime Assessment of Chronic Pain in Youth
Acronym: TRAC-Pain
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Wake Forest University Health Sciences (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Laura E Simons, Professor of Anesthesiology, Perioperative, and Pain Medicine (Pediatric), Stanford University
Other Study IDs: 77005; UG3NS139943 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TRAC-Pain Cohort: For 12 weeks, participants will wear a smartwatch for continuous physiological, sleep, and physical activity monitoring, and complete daily self-reported surveys on pain, mood, and stress. At the end of the study, participants will complete a stress task (Trier Social Stress Task) and a functional task (Sit-to-Stand Test) along with a feedback interview.

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of using wearable digital health technology for continuous monitoring of physiological, sleep, and physical activity data in adolescents with chronic musculoskeletal (MSK) pain. This research aims to develop objective digital endpoints of the pain experience to improve diagnosis, prevention, and treatment outcomes.

DETAILED DESCRIPTION:
Up to 5% of adolescents (~3.5 million in the US alone) suffer from high-impact chronic musculoskeletal (MSK) pain, affecting quality of life, school attendance, mood, and family function, and posing a significant economic burden of $19.5 billion annually in the US. A substantial proportion of these youths continue to suffer from pain into adulthood. Chronic MSK pain is characterized by a complex biological response, including physiological disturbances in cognition, sleep, and energy levels (fatigue), and is associated with impairments in both physical and emotional function. The chronic pain experience fluctuates over time with intra- and inter-daily variations and the occurrence of pain flares, contributing to unpredictability, uncertainty, and greater impairment.

Current gold standard self-report assessments are burdensome and fail to provide comprehensive, reliable measures of the pain experience due to inherent recall bias. A potential solution lies in the widespread adoption of digital health technologies, particularly wearable devices, which offer continuous monitoring of physiological, sleep, and physical activity data. This approach can yield unprecedented insights into individual health, informing diagnosis, prevention, monitoring, and treatment.

Through artificial intelligence (AI) and machine learning (ML), several groundbreaking digital biosignatures of human health have been developed by the research team, including those for glucose variability, preterm birth, panic attacks, fall risk, and surgical recovery. This real-time, personalized approach not only empowers patients but also enables healthcare providers to make more informed decisions, optimizing treatment strategies and improving outcomes. Despite these advancements, less than half of adolescents with chronic MSK pain who undergo pain treatment experience meaningful improvement.

The scientific rationale of this proposal is to overcome the limitations of self-report by integrating precise physiological, sleep, and physical activity measures from wearable devices with AI/ML to develop and validate a monitoring digital biosignature of the individual pain experience in youth with MSK pain. This biosignature will monitor the pain experience, track its progression, assess responses to interventions, and evaluate impacts on quality of life.

The research team is well positioned to execute these aims with: (1) a diverse, highly skilled team with expertise in digital technology, AI/ML, digital endpoint development, and clinical trials, alongside clinical expertise in chronic pain in youth and lived experience from patients, caregivers, and pain advocacy groups; (2) a secure, scalable, centralized, and standardized digital data collection, processing, and storage system; and (3) cutting-edge preliminary data supporting the capability to develop this digital health biosignature.

UG3/Discovery Phase: The research team will enroll up to 500 youth (ages 14-24) with chronic MSK pain, capturing continuous physiological (heart, respiratory), sleep, and physical (activity level, mobility, gait) activity metrics via wearables. Repeated intra-daily self-reports of the pain experience (pain interference, pain intensity, fatigue, mood, stress, pain flares) will be collected over 12 weeks. For a subset, data from physical and social stress tasks will also be gathered. The aim is to assess feasibility and relevance, develop a digital biosignature of the pain experience, and prepare for the UH3 phase through outreach and collaboration. Consultations with individuals with lived experience, those experiencing health disparities, and the FDA will ensure the relevance and acceptability of the biosignature and promote recruitment of underrepresented youth, coupled with scalability for clinical use.

UH3/Validation Phase: The research team will enroll up to 400 diverse youth with chronic MSK pain, capturing wearable and self-reported pain experience metrics over 12 weeks: a 4-week baseline followed by 8 weeks of abnormal reading-triggered alerts. The aim of this phase is to clinically validate the digital biosignature of the pain experience, and evaluate the accuracy and potential of an enhanced wellness alert system.

Significance and Clinical Impact: The successful development and validation of digital endpoints for the pain experience are crucial for advancing pain management. These endpoints promise to improve therapeutic development by providing robust, objective measures of treatment response. The outcomes of this study will be foundational for seeking regulatory approval for the commercialization of the associated software or for disseminating open-source analysis packages for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* The patient has musculoskeletal pain in 1 or more anatomic regions.
* Pain persists for > 3 months.
* Pain is associated with significant distress or life interference.

Exclusion Criteria:

* Significant cognitive impairment (e.g., unable to communicate)
* Hospitalization in the past 30 days for something other than their pain condition
* Currently undergoing treatment for cancer
* Reports only headache, orofacial, or visceral pain
* Currently pregnant or think you might become pregnant in the next 3 months

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 14 - 24 year old adolescents with chronic musculoskeletal pain
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pain, Enjoyment of Life, and General Activity (PEG) Scale | Daily from baseline to discharge, for a duration of 12 weeks
  The PEG scale, a subset of the Brief Pain Inventory (BPI), evaluates pain intensity and its impact on enjoyment of life and general activity using a ranked scale (score 0 = "no interference" to 10 = "highest level of interference") with a higher score reflecting greater disruption in daily functioning.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) of Present Pain | Daily from baseline to discharge, for a duration of 12 weeks
  The Numeric Rating Scale (NRS) for Present pain assesses the intensity of current pain using a ranked scale (0 = "no pain" to 10 = "the worst possible pain") with a higher score reflecting greater pain severity.
Numeric Rating Scale (NRS) Fatigue | Daily from baseline to discharge, for a duration of 12 weeks
  The Numeric Rating Scale (NRS) for Fatigue measures the level of fatigue experienced using a ranked scale (0 = "no fatigue" to 10 = "the most extreme fatigue") with a higher score indicating greater exhaustion.
Numeric Rating Scale (NRS) Stress Level | Daily from baseline to discharge, for a duration of 12 weeks
  The Numeric Rating Scale (NRS) for Stress Level evaluates the severity of stress using a ranked scale (0 = "no stress" to 10 = "the highest level of stress") with a higher score reflecting increased stress intensity.
Numeric Rating Scale (NRS) Activity Level | Daily from baseline to discharge, for a duration of 12 weeks
  The Numeric Rating Scale (NRS) for activity level assesses a person's level of physical activity using a ranked scale (0 = "no activity" to 10 = "the highest possible level of activity") with a higher score reflecting greater engagement in physical activity.
Numeric Rating Scale (NRS) Sleep Quality | Daily from baseline to discharge, for a duration of 12 weeks
  The Numeric Rating Scale (NRS) for Sleep Quality evaluates the quality of sleep using a ranked scale (0 = "the worst possible sleep quality" to 10 = "the best possible sleep quality") with a higher score reflecting better sleep quality.

OTHER OUTCOMES:
Adolescent Sleep Wake Scale - Short Form (ASWS-SF) | Baseline and Discharge (at 12 weeks)
  The Adolescent Sleep Wake Scale - Short Form (ASWS-SF) evaluates sleep patterns and quality in adolescents using a ranked scale (0 = "worst possible sleep quality" to 10 = "best possible sleep quality"), with a higher score reflecting better sleep quality.
Adverse Events | As needed, from baseline to discharge, for a duration of 12 weeks
  The Adverse Events scale monitors for any adverse effects related to the intervention, tracking their frequency and severity, with higher values indicating a greater number or severity of adverse events.
Brief Pain Inventory Short Form (BPI-SF) | Baseline and Discharge (at 12 weeks)
  The Brief Pain Inventory Short Form (BPI-SF) evaluates pain severity and its interference with daily functioning using a 10-point Likert scale (0 = "no pain/interference" to 10 = "worst possible pain/interference"), with a higher score indicating greater pain severity and disruption.
Child Activity Limitations Interview-9 (CALI-9) | Baseline and Discharge (at 12 weeks)
  The Child Activity Limitations Interview-9 (CALI-9) assesses activity limitations due to pain in children and adolescents using a ranked scale (0 = "no activity limitations" to 10 = "unable to engage in any activities"), with a higher score reflecting greater restrictions in daily activities.
Generalized Anxiety Disorder-2 (GAD-2) | Daily from baseline to discharge, for a duration of 12 weeks
  The Generalized Anxiety Disorder-2 (GAD-2) screens for generalized anxiety symptoms using two questions, scored on a scale from 0 to 6 (0 = "no anxiety symptoms" to 6 = "severe anxiety symptoms"), with a higher score indicating greater anxiety severity.
Healthcare Use Diary | As needed, from baseline to discharge, for a duration of 12 weeks
  The Healthcare Use Diary records the frequency and type of healthcare services used, with higher values indicating greater healthcare utilization.
McGill Pain Questionnaire 2 (SF-MPQ-2) | Baseline
  The McGill Pain Questionnaire 2 (SF-MPQ-2) measures the sensory, affective, and evaluative dimensions of pain using a ranked scale (0 = "no pain" to 10 = "worst possible pain"), with a higher score indicating more severe pain experiences.
National Institute on Drug Abuse-2 (NIDA-2) | Baseline and Discharge (at 12 weeks)
  The National Institute on Drug Abuse-2 (NIDA-2) screens for substance use risk and behaviors using a 0 to 6 scale (0 = "no substance use risk" to 6 = "highest substance use risk"), with a higher score indicating increased risk.
Net Promoter Score (NPS) | Discharge (at 12 weeks)
  The Net Promoter Score (NPS) measures the likelihood of recommending the intervention to others using a scale from 0 to 10 (0 = "not at all likely to recommend" to 10 = "extremely likely to recommend"), with a higher score indicating greater satisfaction.
Pain Catastrophizing Scale - Children (PCS-C) | Baseline and Discharge (at 12 weeks)
  The Pain Catastrophizing Scale - Children (PCS-C) assesses negative thoughts and feelings related to pain using six questions, scored from 0 to 24 (0 = "no catastrophizing" to 24 = "highest level of catastrophizing"), with a higher score indicating greater pain-related distress
Pain Flare | As needed, from baseline to discharge, for a duration of 12 weeks
  The Pain Flare scale tracks the occurrence and severity of pain flare-ups using a ranked scale (0 = "no pain flare" to 10 = "worst possible pain flare"), with a higher score reflecting more intense and frequent pain exacerbations
Pain Wellness Behaviors | As needed, from baseline to discharge, for a duration of 12 weeks
  The Pain Wellness and Daily Events scale logs daily wellness activities and notable events that might affect pain levels, providing insight into patterns and triggers.
Pain Wellness and Daily Events | As needed, from baseline to discharge, for a duration of 12 weeks
  The Pain Wellness Behaviors scale assesses engagement in behaviors that promote pain management and overall wellness using a ranked scale (0 = "no engagement in wellness behaviors" to 10 = "consistent engagement in wellness behaviors"), with a higher score reflecting greater adherence to positive health behaviors.
Patient Global Impression of Change (PGIC) | Baseline and Discharge (at 12 weeks)
  The Patient Global Impression of Change (PGIC) measures the patient's overall perception of improvement using a ranked scale (0 = "no improvement" to 10 = "greatest possible improvement"), with a higher score indicating greater perceived positive change.
Patient Health Questionnaire-2 (PHQ-2) | Daily from baseline to discharge, for a duration of 12 weeks
  The Patient Health Questionnaire-2 (PHQ-2) screens for depressive symptoms using two questions, scored from 0 to 6 (0 = "no depressive symptoms" to 6 = "severe depressive symptoms"), with a higher score indicating greater severity of depressive symptoms.
Patient-Reported Outcomes Measurement Information System Fatigue (PROMIS Fatigue) | Baseline and Discharge (at 12 weeks)
  The Patient-Reported Outcomes Measurement Information System Fatigue (PROMIS-Fatigue) evaluates the frequency and intensity of fatigue using a ranked scale (0 = "no fatigue" to 10 = "most severe fatigue"), with a higher score indicating greater fatigue severity.
Patient-Reported Outcomes Measurement Information System Physical Function Short Form 8c (PROMIS Physical Function) | Baseline and Discharge (at 12 weeks)
  The Patient-Reported Outcomes Measurement Information System Physical Function Short Form 8c (PROMIS Physical Function) measures physical functioning capabilities and limitations using a ranked scale (0 = "severe limitations" to 10 = "no limitations"), with a higher score indicating better physical function.
Patient-Reported Outcomes Measurement Information System Stress Experiences Short Form 4a (PROMIS Stress) | Baseline and Discharge (at 12 weeks)
  The Patient-Reported Outcomes Measurement Information System Stress Experiences Short Form 4a (PROMIS Stress) assesses perceived stress levels over the past seven days using a ranked scale (0 = "no stress" to 10 = "highest level of stress"), with a higher score indicating greater stress.
Positive and Negative Affect Schedule - 10 Item (PANAS-10) | Daily from baseline to discharge, for a duration of 12 weeks
  The Positive and Negative Affect Schedule - 10 Item (PANAS-10) measures both positive and negative affect using ten items, scored separately from 0 to 50 (0 = "no affect" to 50 = "highest affect intensity"), with a higher score reflecting greater emotional intensity.
Social Determinants of Health (SDOH) | Baseline
  The Social Determinants of Health (SDOH) scale assesses factors such as socioeconomic status, education, and environment that influence health outcomes, with a higher score indicating greater social risk factors.
Theoretical framework of acceptability (TFA) | Discharge (at 12 weeks)
  The Theoretical Framework of Acceptability (TFA) scale evaluates participant perceptions of an intervention's acceptability using a ranked scale (0 = "not acceptable" to 10 = "highly acceptable"), with a higher score reflecting greater acceptance and perceived usefulness.
Usage metrics | Daily from baseline to discharge, for a duration of 12 weeks
  The Usage Metrics scale assesses participant engagement with the intervention by tracking hours of smartwatch wear, percentage of completed surveys, and check-ins, with higher values indicating greater adherence and participation.
World Health Organization Quality of Life 2 Item (WHOQOL-2) | Baseline and Discharge (at 12 weeks)
  The World Health Organization Quality of Life 2 Item (WHOQOL-2) measures overall quality of life and general health using a ranked scale (0 = "worst quality of life" to 10 = "best quality of life"), with a higher score indicating better quality of life and health perception.
Pediatric Pain Screening Tool (PPST) | Baseline and discharge (at 12 weeks)
  The Pediatric Pain Screening Tool (PPST) is a 9-item self-report measure designed to assess both physical and psychosocial aspects of pain in youth

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Robust individual level data will be available to share, not just group level data.